CLINICAL TRIAL: NCT03192410
Title: Prospective Cohort Study of 4,837 Post-myocardial Infarction Patients (Alpha Omega Cohort)
Status: Active, not recruiting | Type: Observational
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Geleijnse, Professor of Nutrition and Cardiovascular Disease, Wageningen University
Other Study IDs: Alpha Omega Cohort
Record Dates: First submitted 2017-06-10; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Cardiovascular Diseases; Mortality; Type 2 Diabetes Mellitus; Cognitive Decline; Mental Well-being; Kidney Function
Keywords: myocardial infarction; cardiovascular diseases; mortality; post-myocardial infarction patients; risk prediction; kidney function; mental well-being; cardiovascular drug treatment
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Cognitive Dysfunction; Psychological Well-Being; Myocardial Infarction | interventions — Eating; Health; DNA; Mental Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Non-fasting venous blood samples were taken in 4785 patients at baseline, in 810 patients after 20 months and in 2503 patients after 40 months of follow-up. DNA has been extracted for genotyping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Dietary intake — Intake of nutrients, foods, food groups, beverages; dietary patterns.
Behavioral: Lifestyle factors — Physical activity; smoking; alcohol use; educational level.
Biological: Blood biomarkers — Biomarkers of dietary intake (e.g. fatty acids); biomarkers of disease.
Biological: Health — Current health status; medical history; medication use; self-rated health; risk factors for disease (e.g. body mass index, blood pressure, blood lipids, glucose)
Genetic: DNA — SNPs (GWAS)
Biological: Mental well-being — Cognitive function; dispositional optimism; depression.

SUMMARY:
The Alpha Omega Cohort is a prospective study of 4,837 state-of-the-art drug-treated Dutch patients aged 60-80 years who had a clinically diagnosed myocardial infarction up to 10 years before enrolment. During the first 40 months of follow-up, patients took part in an experimental study of low doses n-3 fatty acids (Alpha Omega Trial, ClinicalTrials.gov NCT00127452). At baseline (2002-2006), data on medical history, medication use, diet, lifestyle and other factors were collected by means of questionnaires. Patients were physically examined by trained research nurses and blood samples were obtained. Follow-up for vital status and cause-specific mortality is ongoing. The trial was approved by a central medical ethics committee (Haga Hospital, The Hague, The Netherlands) and all patients provided written informed consent.

DETAILED DESCRIPTION:
Details are reported in publications.

ELIGIBILITY:
The Alpha Omega Cohort is a prospective cohort study. The cohort originated from the Alpha Omega Trial, a 40-month intervention study of low doses of n-3 fatty acids (in margarine spreads) and cardiovascular events (NCT00127452). The in/exclusion criteria were defined for the Alpha Omega Trial.

Inclusion criteria:

* Men and women
* Aged 60 through 80 y
* Verified clinically diagnosed myocardial infarction up to 10 y before entry into the study
* Written informed consent

Exclusion criteria:

* Living in a nursing home or other institution
* Participation in another scientific study
* Habitual margarine intake < 10 g per day
* Habitual fish intake > 150 g per day
* Habitual alcohol intake > 6 drinks per day
* Use of fish oil capsules or other supplements containing omega-3 fatty acids
* Presence of cancer with < 1 y of life expectancy
* Cognitive impairment, as indicated by the Mini Mental State Examination (score <= 21)
* Unintended weight loss > 5 kg in the past year
* Lack of facilities for cooled margarine storage at home
* Inability or unwillingness to comply with study procedures

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 4837 patients (78% male) with a history of myocardial infarction up to 10 y before entry into the study, recruited from 32 hospitals in the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 4837 (Actual)
Dates: Start 2002-04 (Actual); Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality | From entry into the study (baseline: 2002-2006) through study completion
  Death from cardiovascular disease, obtained from causes of death register of Statistics Netherlands
All-cause mortality | From entry into the study (baseline: 2002-2006) through study completion
  Vital status obtained from municipal population registers in the Netherlands
Major cardiovascular events | From entry into the study (baseline: 2002-2006) until November 2009
  Incidence of fatal and nonfatal cardiovascular events and hospitalisations for cardiac interventions, based on verified information from GP records, hospital records and mortality registers

SECONDARY OUTCOMES:
Coronary heart disease | From entry into the study (baseline: 2002-2006) through study completion
  Incidence of fatal and non-fatal coronary heart disease, based on verified information from GP records, hospital records and mortality registers
Stroke | From entry into the study (baseline: 2002-2006) through study completion
  Incidence of fatal and non-fatal stroke, based on verified information from GP records, hospital records and mortality registers
Non-cardiovascular mortality | From entry into the study (baseline: 2002-2006) through study completion
  Death from cancer or other non-cardiovascular causes, obtained from causes of death register of Statistics Netherlands
Type 2 diabetes | From entry into the study (baseline: 2002-2006) until November 2009
  Incidence of type 2 diabetes, on basis of self-reported physician diagnosis, use of antidiabetic drugs, or elevated blood glucose
Kidney function | From entry into the study (baseline: 2002-2006) until November 2009
  Change in serum cystatin C-based estimated glomerular filtration rate
Cognitive function | From entry into the study (baseline: 2002-2006) until November 2009
  Change in global cognitive function, based on Mini Mental State Examination (MMSE) score

OTHER OUTCOMES:
Depression | After 40 months of follow-up
  Score on 15-item Geriatric Depression Scale
Dispositional optimism | After 40 months of follow-up
  Scores on a 4-item questionnaire and the (revised) Life Orientation Test (LOT-R)
Body weight | From entry into the study (baseline: 2002-2006) until November 2009
  Change in body weight, assessed by trained research nurses
Blood pressure | From entry into the study (baseline: 2002-2006) until November 2009
  Change in office blood pressure, assessed by trained research nurses
Blood lipids | From entry into the study (baseline: 2002-2006) until November 2009
  Change in non-fasting serum total, LDL and HDL cholesterol, assessed by standard laboratory methods
Glucose metabolism | From entry into the study (baseline: 2002-2006) until November 2009
  Change in non-fasting plasma glucose, insulin and HbA1C, assessed by standard laboratory methods
DNA genotype | At baseline (2002-2006)
  DNA genotype, assessed by Global Screening Array (Illumina, Inc.)
Biochemical markers of Inflammation | From entry into the study (baseline: 2002-2006) until November 2009
  Change in blood biomarkers of inflammation, assessed by MesoScale assays
Biochemical markers of endothelial function | From entry into the study (baseline: 2002-2006) until November 2009
  Change in blood biomarkers of endothelial function, assessed by MesoScale assays
Biomarkers of cardiac function | From entry into the study (baseline: 2002-2006) until November 2009
  Change in blood biomarkers of cardiac function (e.g, NT-proBNP, troponin), assessed by chemiluminescence
Biomarkers of kidney function | From entry into the study (baseline: 2002-2006) until November 2009
  Change in blood biomarkers of kidney function, assessed by immunoassay
Prostate-specific antigen (PSA) | From entry into the study (baseline: 2002-2006) until November 2009
  Change in blood total PSA concentration, assessed by immunometric assay
Testosterone | From entry into the study (baseline: 2002-2006) until November 2009
  Change in serum testosterone concentration, assessed by immunoassay
Circulating fatty acids | From entry into the study (baseline: 2002-2006) until November 2009
  Change in concentration of fatty acids (percent weight) in plasma cholesteryl esters

CONTACTS AND LOCATIONS:
Overall Officials: Johanna M Geleijnse, PhD, Principal Investigator — Wageningen University, Division of Human Nutrition
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Geleijnse JM, Giltay EJ, Schouten EG, de Goede J, Oude Griep LM, Teitsma-Jansen AM, Katan MB, Kromhout D; Alpha Omega Trial Group. Effect of low doses of n-3 fatty acids on cardiovascular diseases in 4,837 post-myocardial infarction patients: design and baseline characteristics of the Alpha Omega Trial. Am Heart J. 2010 Apr;159(4):539-546.e2. doi: 10.1016/j.ahj.2009.12.033. PMID 20362710
- [Result] Kromhout D, Giltay EJ, Geleijnse JM; Alpha Omega Trial Group. n-3 fatty acids and cardiovascular events after myocardial infarction. N Engl J Med. 2010 Nov 18;363(21):2015-26. doi: 10.1056/NEJMoa1003603. Epub 2010 Aug 28. PMID 20929341
- [Result] Sijtsma FP, Soedamah-Muthu SS, de Goede J, Oude Griep LM, Geleijnse JM, Giltay EJ, de Boer MJ, Jacobs DR Jr, Kromhout D. Healthy eating and lower mortality risk in a large cohort of cardiac patients who received state-of-the-art drug treatment. Am J Clin Nutr. 2015 Dec;102(6):1527-33. doi: 10.3945/ajcn.115.112276. Epub 2015 Oct 21. PMID 26490494
- [Result] Hoogeveen EK, Geleijnse JM, Kromhout D, Stijnen T, Gemen EF, Kusters R, Giltay EJ. Effect of omega-3 fatty acids on kidney function after myocardial infarction: the Alpha Omega Trial. Clin J Am Soc Nephrol. 2014 Oct 7;9(10):1676-83. doi: 10.2215/CJN.10441013. Epub 2014 Aug 7. PMID 25104273
- [Result] Soedamah-Muthu SS, Geleijnse JM, Giltay EJ, Kromhout D; Alpha Omega Trial Group. Cardiovascular risk factor management of myocardial infarction patients with and without diabetes in the Netherlands between 2002 and 2006: a cross-sectional analysis of baseline data. BMJ Open. 2012 Oct 31;2(6):e001360. doi: 10.1136/bmjopen-2012-001360. Print 2012. PMID 23117562
- [Result] Soedamah-Muthu SS, Geleijnse JM, Giltay EJ, de Goede J, Oude Griep LM, Waterham E, Teitsma-Jansen AM, Mulder BJ, de Boer MJ, Deckers JW, Zock PL, Kromhout D; for the Alpha Omega Trial Group. Levels and trends in cardiovascular risk factors and drug treatment in 4837 elderly Dutch myocardial infarction patients between 2002 and 2006. Neth Heart J. 2012 Feb 8;20(3):102-9. doi: 10.1007/s12471-012-0248-z. Online ahead of print. PMID 22314614
- [Derived] Evers I, Cruijsen E, Kornaat I, Winkels RM, Busstra MC, Geleijnse JM. Dietary magnesium and risk of cardiovascular and all-cause mortality after myocardial infarction: A prospective analysis in the Alpha Omega Cohort. Front Cardiovasc Med. 2022 Aug 12;9:936772. doi: 10.3389/fcvm.2022.936772. eCollection 2022. PMID 36035961
- [Derived] Cruijsen E, Indyk IM, Simon AWE, Busstra MC, Geleijnse JM. Potato Consumption and Risk of Cardiovascular Mortality and Type 2 Diabetes After Myocardial Infarction: A Prospective Analysis in the Alpha Omega Cohort. Front Nutr. 2022 Jan 27;8:813851. doi: 10.3389/fnut.2021.813851. eCollection 2021. PMID 35155529
- [Derived] Pertiwi K, Kupers LK, de Goede J, Zock PL, Kromhout D, Geleijnse JM. Dietary and Circulating Long-Chain Omega-3 Polyunsaturated Fatty Acids and Mortality Risk After Myocardial Infarction: A Long-Term Follow-Up of the Alpha Omega Cohort. J Am Heart Assoc. 2021 Dec 7;10(23):e022617. doi: 10.1161/JAHA.121.022617. Epub 2021 Nov 30. PMID 34845924
- [Derived] Cruijsen E, de Ruiter AJ, Kupers LK, Busstra MC, Geleijnse JM. Alcohol intake and long-term mortality risk after myocardial infarction in the Alpha Omega Cohort. Am J Clin Nutr. 2022 Mar 4;115(3):633-642. doi: 10.1093/ajcn/nqab366. PMID 34734223
- [Derived] Cruijsen E, Jacobo Cejudo MG, Kupers LK, Busstra MC, Geleijnse JM. Dairy consumption and mortality after myocardial infarction: a prospective analysis in the Alpha Omega Cohort. Am J Clin Nutr. 2021 Jul 1;114(1):59-69. doi: 10.1093/ajcn/nqab026. PMID 33826695
- [Derived] van Westing AC, Eckl MR, Kupers LK, Pertiwi K, Hoogeveen EK, Geleijnse JM. Plasma fatty acids and kidney function decline in post-myocardial infarction patients of the Alpha Omega Cohort. Nutr Metab Cardiovasc Dis. 2021 May 6;31(5):1467-1476. doi: 10.1016/j.numecd.2021.01.012. Epub 2021 Jan 29. PMID 33744039
- [Derived] Esmeijer K, Geleijnse JM, Giltay EJ, Stijnen T, Dekker FW, de Fijter JW, Kromhout D, Hoogeveen EK. Body-fat indicators and kidney function decline in older post-myocardial infarction patients: The Alpha Omega Cohort Study. Eur J Prev Cardiol. 2018 Jan;25(1):90-99. doi: 10.1177/2047487317739986. Epub 2017 Nov 2. PMID 29095051
- [Derived] Rius-Ottenheim N, Kromhout D, Sijtsma FPC, Geleijnse JM, Giltay EJ. Dietary patterns and mental health after myocardial infarction. PLoS One. 2017 Oct 16;12(10):e0186368. doi: 10.1371/journal.pone.0186368. eCollection 2017. PMID 29036212
- [Derived] van Dongen LH, Molenberg FJ, Soedamah-Muthu SS, Kromhout D, Geleijnse JM. Coffee consumption after myocardial infarction and risk of cardiovascular mortality: a prospective analysis in the Alpha Omega Cohort. Am J Clin Nutr. 2017 Oct;106(4):1113-1120. doi: 10.3945/ajcn.117.153338. Epub 2017 Aug 23. PMID 28835365
- [Derived] Molenberg FJM, de Goede J, Wanders AJ, Zock PL, Kromhout D, Geleijnse JM. Dietary fatty acid intake after myocardial infarction: a theoretical substitution analysis of the Alpha Omega Cohort. Am J Clin Nutr. 2017 Sep 1;106(3):895-901. doi: 10.3945/ajcn.117.157826. PMID 28793994
- See also: Website of the Alpha Omega Trial (experimental phase of Alpha Omega Cohort) — http://www.alphaomegatrial.com